CLINICAL TRIAL: NCT00331279
Title: The Effect of Cinnamon Extract on Insulin Resistance Parameters in Polycystic Ovary Syndrome: A Pilot Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency); Integrity Neutraceuticals, Inc. Sarasota, FL (Industry)
Responsible Party: Principal Investigator, Rogerio A. Lobo, Professor, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AAAA8837
Record Dates: First submitted 2006-05-25; First posted 2006-05-29 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2011-01

CONDITIONS: Polycystic Ovary Syndrome
Keywords: polycystic ovary syndrome; insulin resistance; cinnamon
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cinnamon Extract (Active Comparator): A purified aqueous abstract of cinnamon in a 500mg tablet will be taken by each patient before lunch and dinner, making a total of one gram per day for eight weeks.
  Interventions: Drug: Oral Cinnamon Extract
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral Cinnamon Extract — A purified aqueous abstract of cinnamon in a 500mg tablet will be taken by each patient before lunch and dinner, making a total of one gram per day for eight weeks.
  Other Names: Cinnamon Extract
  Arms: Cinnamon Extract
Drug: Placebo — Placebo pills in likeness of the cinnamon extract
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether oral cinnamon extract are effective in reducing insulin resistance parameters in women with polycystic ovary syndrome.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is a very common condition found in women of childbearing age. PCOS patients often have irregular periods, extra hair growth, or difficulty becoming pregnant. The syndrome can also be associated with more serious conditions such as heart disease, diabetes, or cancer of the uterus.

Although no one knows the cause of the syndrome, scientific studies showed that having too much insulin can be one of the reasons. In fact, almost every overweight woman with PCOS has been found to have high insulin levels.

Medications that lower the body's insulin level used to treat people with diabetes mellitus have also been used very successfully to treat some of the symptoms of PCOS such as irregular periods.

Recently studies using rats and mice have shown that a commonly used spice, cinnamon, may also reduce the body's insulin level. Another study showed that daily use of cinnamon for forty days lowered the blood sugar level in patients with diabetes. The purpose of this study is to see if cinnamon can lower the insulin level in women with PCOS. If so, it can also be used as a treatment for irregular periods as well.

Half of the patients in the study will take premade cinnamon extract pills twice a day while the other half will take placebo pills (pills with no cinnamon extract) twice a day for eight weeks. Blood tests measuring insulin, substances important for insulin action, cholesterol, and glucose (sugar) will be taken before and after the eight weeks of medication. A total of three separate visits will be needed to finish the study. At the end of the study, we will then compare the blood glucose, insulin, and cholesterol levels between the patients that took cinnamon and the patients that took placebo.

ELIGIBILITY:
Inclusion Criteria:

* Polycystic ovary syndrome

Exclusion Criteria:

* Diabetes mellitus, hyperprolactinemia, thyroid disorders, and hypertension

Ages: 23 Years to 47 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2005-08; Primary Completion 2005-09 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Fasting glucose | Duration of study
Fasting insulin | Duration of study
HOMA-IR | Up to 8 weeks after treatment
QUICKI | Up to 8 weeks after treatment
Insulin sensitivity index (Matsuda) | Up to 8 weeks after treatment

SECONDARY OUTCOMES:
Total testosterone | Up to 8 weeks after treatment
Sex hormbone binding globulin | Up to 8 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Rogerio Lobo, M.D., Principal Investigator — Columbia University
Locations (1):
- Center for Women's Reproductive Care, New York, New York, United States